CLINICAL TRIAL: NCT06813079
Title: ADOPT: Adaptive Organoid-Based Precision Therapy Study in Pancreatic Cancer - A Prospective Single-Arm Phase II Trial
Brief Title: Using Tumor Models to Determine Treatments
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADOPT; 24-5059 (Other: University Health Network)
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Ductal Carcinoma; Advanced Cancer; Epithelial Tumor
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Carcinoma | interventions — cobimetinib; ponatinib; brigatinib; Colchicine; selinexor; abemaciclib; neratinib; Doxorubicin; Etoposide; ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Patients in this cohort will be entering the study for treatment for progressive disease.
  Interventions: Drug: Cobimetinib; Drug: Ponatinib; Drug: Brigatinib; Drug: Colchicine; Drug: Selinexor; Drug: Abemaciclib; Drug: Neratinib; Drug: Doxorubicin; Drug: Etoposide; Drug: Ceritinib
- Cohort B (Experimental): Patients in this cohort will be entering the study for maintenance therapy with stable disease.
  Interventions: Drug: Cobimetinib; Drug: Ponatinib; Drug: Brigatinib; Drug: Colchicine; Drug: Selinexor; Drug: Abemaciclib; Drug: Neratinib; Drug: Doxorubicin; Drug: Etoposide; Drug: Ceritinib

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib is an antineoplastic agent and selective inhibitor of the mitogen-activated extracellular kinase (MEK) pathway.
  Participants will take cobimetinib by mouth (orally), once a day on days 1 to 21 followed by a 7-day break of each cycle. A cycle will be 28 days in length.
Drug: Ponatinib — Ponatinib is a type of drug called a protein tyrosine kinase inhibitor (TKI). Tyrosine kinases are proteins that act as chemical messengers to stimulate cancer cells to grow. Ponatinib blocks and interferes with a number of protein kinases. It is called a multi kinase inhibitor.
  Participants will take ponatinib by mouth (orally), once a day, every day of each cycle. A cycle will be 28 days.
Drug: Brigatinib — Brigatinib is a type of cancer growth blockers called a tyrosine kinase inhibitor (TKI). It blocks chemical signals (enzymes) from tyrosine kinase proteins. Tyrosine kinases help to send growth signals in cells, so blocking them stops the cell growing and dividing.
  Participants will take brigatinib by mouth (orally), once a day for the first 7 days. If participants are able to tolerate the dose during the first 7 days, they will take the doubled dose orally, once a day until end of the cycle (day 8 to day 28). Each cycle will be 28 days in length.
Drug: Colchicine — Colchicine is an alkaloid that affects the way the body responds to uric acid crystals, and reduces swelling and pain.
  On the first day, participants will take two tablets of colchicine by mouth (orally), then one tablet orally one hour later. Starting the second day, participants will take one tablet of colchicine once or twice a day, every day of each cycle. A cycle will be 28 days in length. The study doctor will decide whether participants will take colchicine once or twice a day.
Drug: Selinexor — Selinexor blocks a protein called CRM1, a protein within the cell, and may help keep cancer cells from growing and may kill them. It is a type of small molecule inhibitor.
  Participants will take selinexor by mouth (orally), once a week on days 1, 8, 15, and 22 of each cycle. A cycle will be 28 days in length.
Drug: Abemaciclib — Abemaciclib belongs to a class of medications called kinase inhibitors. Abemaciclib works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells.
  Participants will take abemaciclib by mouth (orally), twice a day, every day of each cycle. A cycle will be 28 days in length.
Drug: Neratinib — Neratinib is a targeted cancer drug that works on a protein called human epidermal growth factor receptor 2 (HER2). HER2 proteins make cells divide and grow. Some cancers have large amounts of HER2 proteins which can cause cancer cells to divide and grow faster. Neratinib works by locking onto the HER2 on the cancer cells. So it stops the cells from growing.
  Participants will take neratinib by mouth (orally), once a day, every day of each cycle. Dose will increase weekly, until week 3. On week 3 and onward, participants will take the same dose. A cycle will be 28 days in length.
Drug: Doxorubicin — Doxorubicin is a type of chemotherapy drug called an anthracycline. It slows or stops the growth of cancer cells by blocking an enzyme called topo isomerase 2. Cancer cells need this enzyme to divide and grow.
  Participants will receive doxorubicin by vein (intravenous infusion or IV) in clinic, over 60-90 minutes, once every cycle. A cycle will be 21 days in length. Participants may receive 6-8 cycles of study drug.
Drug: Etoposide — Etoposide is a chemotherapy drug that destroys quickly dividing cells, such as cancer cells.
  Participants will receive etoposide by mouth (orally), twice a day, on days 1 to 7 of every cycle. On days 8 to 21, there will be no dosing. A cycle will be 21 days in length.
Drug: Ceritinib — Ceritinib is a tyrosine kinase inhibitor. It works by blocking an enzyme called anaplastic lymphoma kinase (ALK). Ceritinib only works in cancer cells that have an overactive version of ALK.
  Participants will take ceritinib by mouth (orally), once a day, every day of each cycle. A cycle will be 28 days in length.

SUMMARY:
The purpose of this study is to see if using Patient Derived Organoids (PDO) to choose a drug for the treatment of pancreatic cancer individually for each patient is useful. The study will look at the number of participants who have a response to their assigned drug.

DETAILED DESCRIPTION:
PDO is a three-dimensional experimental model grown in a laboratory from patient's tumour tissues. PDO is used to test different drugs and select the drugs that may work for treating the patient's cancer. Researchers will review participants' PDO drug results from other studies from which they participated in and will identify the drug that seem to have the best effect on the PDO model. Participants will be offered to receive that drug during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over
2. Ability to understand and willing to sign a written informed consent form in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to screening to document their willingness to participate.
3. Advanced inoperable malignant epithelial pancreatic ductal carcinomas (i.e. primary diagnosis of ductal adenocarcinoma or acinar cell adenocarcinoma, inclusive of all subtypes)
4. Treatment history meeting one of either:

   1. Stable disease or partial response to FOLFIRINOX (leucovorin calcium/folinic acid, fluorouracil, irinotecan hydrochloride, and oxaliplatin) after at least eight cycles of treatment (Cohort B)
   2. Progression of disease after receiving standard of care chemotherapies (Cohort A).

   i. There is no maximum number of prior lines

   ii. Patients with recurrence within six months of adjuvant-intent chemotherapy will be eligible
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
6. Life Expectancy of greater than 12 weeks
7. Patients must have acceptable organ function
8. Patients must have baseline hepatitis B screening. If they have a positive surface antigen the case will discussed with the hepatologist to determine if therapy is indicated. This does not exclude them from study.
9. Patients must agree to use effective contraceptive methods for the period required by the study.
10. Patients must have measurable disease
11. Patient-derived organoid is sensitive to a drug listed for this study, defined by

    1. Consensus agreement in molecular tumor boards, considering the totality of the genomic and organoid data, and the safety profile of the drug, and the clinical situation
    2. Sensitivity to a drug chosen for the study, based on

    i. IC50 < Cmax (maximum plasma concentration) ii. Area under the curve (AUC) < 30th percentile of cohort iii. Individual assay fulfills quality control metrics c. Matched clinical scenario (maintenance versus treatment) as outlined in this protocol.
12. Able to swallow and tolerate oral medication (as applicable)

Exclusion Criteria:

1. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
2. Patient received last dose of chemotherapy within 21 days prior to Cycle 1 Day 1.
3. Patients with ongoing toxicity ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 2, other than peripheral neuropathy, related to prior anti-tumour treatment.
4. Patients with ongoing peripheral neuropathy of ≥ CTCAE grade 3 will be excluded.
5. Patients concurrently receiving any other anti-cancer therapy (cytotoxic, biologic, radiation, or hormonal other than for replacement) except for medications that are prescribed for supportive care but may potentially have an anti-cancer effect (e.g. megestrol acetate, bisphosphonates). These medications must have been started ≥ one month prior to enrolment in this study.
6. Patients with a history of a severe allergic reaction attributed to compounds of similar or biologic composition to the PDO matched drug may be excluded if assessed by the investigator and determined to be unsafe to proceed.
7. Patients may be on warfarin, low molecular weight heparin or direct factor Xa inhibitors, unless such therapies are prohibited by drug-specific ineligibility criteria.
8. Patients with known active progressive brain metastases. Patients with previously treated brain metastases are eligible, provided that the patient has not experienced a seizure or had a clinically significant change in neurological status within one month prior to screening. All patients with previously treated brain metastases must be stable (clinically and radiologically) for at least one month after completion of treatment and either off steroid treatment or only taking physiological doses of steroids prior to the screening step.
9. Patients with clinically significant pre-existing cardiac conditions, including uncontrolled or symptomatic angina, uncontrolled atrial or ventricular arrhythmias, or symptomatic congestive heart failure.
10. Patients with known left ventricular ejection fraction (LVEF) < 40 % as determined by a multigated acquisition (MUGA) scan or echocardiogram.
11. Patients with stroke (including TIA) or acute myocardial infarction within three months prior to the screening step.
12. Patients with acute gastrointestinal bleeding within one month prior to the screening step.
13. Patients with any other clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements including, but not limited to ongoing or active infection, significant uncontrolled hypertension, or severe psychiatric illness/social situations.
14. Lactating and nursing women.
15. Patients who do not meet drug-specific eligibility requirements for the drug selected by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2028-02-17 (Estimated); Study Completion 2028-02-17 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 3 years

SECONDARY OUTCOMES:
Disease control rate (DCR) | 3 years
Duration of response (DOR) | 3 years
Progression free survival (PFS) | 3 years
Overall survival (OS) | 3 years
Number of side effects experienced with participants in Cohort A assigned to cobimetinib | 3 years
Number of side effects experienced with participants in Cohort B assigned to cobimetinib | 3 years
Number of side effects experienced with participants in Cohort A assigned to ponatinib | 3 years
Number of side effects experienced with participants in Cohort B assigned to ponatinib | 3 years
Number of side effects experienced with participants in Cohort A assigned to brigatinib | 3 years
Number of side effects experienced with participants in Cohort B assigned to brigatinib | 3 years
Number of side effects experienced with participants in Cohort A assigned to colchicine | 3 years
Number of side effects experienced with participants in Cohort B assigned to colchicine | 3 years
Number of side effects experienced with participants in Cohort A assigned to selinexor | 3 years
Number of side effects experienced with participants in Cohort B assigned to selinexor | 3 years
Number of side effects experienced with participants in Cohort A assigned to ceritinib | 3 years
Number of side effects experienced with participants in Cohort B assigned to ceritinib | 3 years
Number of side effects experienced with participants in Cohort A assigned to abemaciclib | 3 years
Number of side effects experienced with participants in Cohort B assigned to abemaciclib | 3 years
Number of side effects experienced with participants in Cohort A assigned to neratinib | 3 years
Number of side effects experienced with participants in Cohort B assigned to neratinib | 3 years
Number of side effects experienced with participants in Cohort A assigned to doxorubicin | 3 years
Number of side effects experienced with participants in Cohort B assigned to doxorubicin | 3 years
Number of side effects experienced with participants in Cohort A assigned to etoposide | 3 years
Number of side effects experienced with participants in Cohort B assigned to etoposide | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Grant, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada